CLINICAL TRIAL: NCT01864993
Title: Glutox Trial. Symptomatic Response to Gluten Challenge in Patients With Suspected Non Celiac Gluten Sensitivity: a Double Blind Crossover Controlled Trial
Brief Title: Symptomatic Response to Gluten Challenge in Patients With Suspected Non Celiac Gluten Sensitivity
Acronym: Glutox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Elli, researcher, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1876/2012; 1876 (Other: Fondazione IRCCS Cà Granda)
Record Dates: First submitted 2013-05-19; First posted 2013-05-30 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Non Celiac Gluten Sensitivity
Keywords: non celiac gluten sensitivity; gluten; irritable bowel syndrome; functional disorders
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- suspected NC gluten sensitive subjects (Experimental): Patients referring gastrointestinal functional disorders will be selected and they will follow a gluten free diet
  Interventions: Dietary Supplement: gluten; Dietary Supplement: Placebo
- suspected NC gluten sensitive (Experimental): Patients referring gastrointestinal functional disorders will be selected and they will follow a gluten free diet
  Interventions: Dietary Supplement: gluten; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: gluten — The enrolled patients will be invited to follow a gluten free diet. Patients responsive to the diet will be invited to assume gluten or placebo following a double blind with cross over scheme
Dietary Supplement: Placebo — Patients responsive to the diet will be invited to blindly assume gluten or placebo following a double blind with cross over scheme

SUMMARY:
Non Celiac Gluten Sensitivity (NCGS) is an emergent syndrome mainly inducing gastrointestinal symptoms. NCGS is suspected to be present in the 6% of the population and thus it represents an important issue in health care. Actually it remains difficult to diagnose and prove due to the lack of established criteria. The investigators intention is to establish a diagnostic flowchart to evaluate the real impact of NCGS in a cohort of patients suffering from functional gastrointestinal symptoms.

DETAILED DESCRIPTION:
The proposed study has been designed to be a randomised double-blind multicenter clinical trial with crossover. The Coordinating Center will be the "Centro per la Prevenzione e la Diagnosi della Malattia Celiaca", Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milano. Secondary enrollment centers will be Italian Gastroenterology Units with outpatient services. Enrollment criteria will be diagnosis of irritable bowel syndrome (IBS) or functional dyspepsia. Patients with other functional gastrointestinal disorders will be included in the group "Functional non specific gastrointestinal symptoms".

After they give their written informed consent, patients will undergo the diagnostic work-up recommended in case of suspected irritable bowel symptoms/functional dyspepsia and aimed at the exclusion of CD or allergy to alimentary antigens by means of serological testing (anti transglutaminase antibodies) or skin tests, or other gastrointestinal diseases. Endoscopic, histologic and/or imaging exams together with supplemental blood tests will be prescribed on individual cases and according with the international guidelines.

Enrolled subjects will be asked to fill

* a checklist for the evaluation of the psychological profile (SCL90 questionnaire, with the particular aim of evaluating levels of anxiety, depression and somatisation);
* a questionnaire about the perceived level of physical and mental health (SF36 questionnaire);
* Ten centimeters long visual analogue scales (VAS) on the level of satisfaction with their health status and on the intensity of the single symptoms.

At the end of the present phase patients will start a GFD for the subsequent three weeks.

At the end of the GFD period patients will fill VAS and SF36. Only those patients presenting a 30% increase of the global VAS score ("GFD Responders") will continue the study. Conversely, non responders will be considered "non gluten sensitive" and they will finish the trial.

Responders to the GFD period will entry the randomisation phase and will undergo a double-blind stimulation test with cross over. Patients will be randomised to assume gluten or placebo for 7 days. After the treatment patients will fill VAS and SF36.

A diagnosis of NCGS will be ascertained in case of symptomatic response limited to gluten ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with gastrointestinal functional disorders (irritable bowel syndrome, functional dyspepsia or unspecified functional gastrointestinal symptoms)

Exclusion Criteria:

* Celiac disease
* Alimentary allergies
* Inflammatory bowel disease
* Major abdominal surgery
* Psychiatric disorders
* Neoplasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analogue Scales | 28 days
  Symptomatic resolution after the instauration of a gluten free diet will be verified by means of VAS scales

SECONDARY OUTCOMES:
Quality of Life | 28 days
  patients with non celiac gluten sensitivity will be evaluated by means of SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, MD, PhD, Principal Investigator — Center for Prevention and Diagnosis of Celiac Disease, Fondazione IRCCS Cà Granda
Locations (5):
- Italy (5):
  - Ospedale Maggiore di Crema, Crema, Italy
  - Ospedale S. Maria, Feltre, Italy
  - Ospedale Di Busto Arsizio, Busto Arsizio, Lombardy
  - Ospedale Valduce di Como, Como, Lombardy
  - Arcispedale S. Maria Nuova, Reggio Emilia

REFERENCES:
- [Derived] Scricciolo A, Lombardo V, Elli L, Bascunan KA, Doneda L, Rinaldi F, Pinto D, Araya M, Costantino A, Vecchi M, Roncoroni L. Use of a proline-specific endopeptidase to reintroduce gluten in patients with non-coeliac gluten sensitivity: A randomized trial. Clin Nutr. 2022 Sep;41(9):2025-2030. doi: 10.1016/j.clnu.2022.07.029. Epub 2022 Jul 31. PMID 35973395